CLINICAL TRIAL: NCT00518778
Title: Fusariosis in Solid-Organ Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Adarsh Bhimrah, UPMC
Other Study IDs: PRO07070159; investigator funding (Other: UPMC)
Record Dates: First submitted 2007-08-17; First posted 2007-08-21 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Solid Organ Transplant; Fusariosis
Keywords: fusariosis; solid organ transplants
MeSH Terms: conditions — Fusariosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This exempt chart review study will try to determine the clinical presentation, prognostic factors, response to different treatment modalities and mortality among patients diagnosed with fusariosis after solid-organ transplantation.

DETAILED DESCRIPTION:
This exempt chart review study will try to determine the clinical presentation, prognostic factors, response to different treatment modalities and mortality among patients diagnosed with fusariosis after solid-organ transplantation.This will help determine prognostic factors, response to different treatment modalities and mortality among patients diagnosed with fusariosis after solid-organ transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Solid-organ transplants (liver, kidney, lung, heart, pancreas, small bowel transplant) diagnosed with fusariosis or infections due to Fusarium, species in our institution

Exclusion Criteria:

* Those subjects that do not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Solid organ transplant patients diagnosed with fusariosis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-08; Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adarsh Bhimraj, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States